CLINICAL TRIAL: NCT07120672
Title: The Role of Peripheral Perfusion Index as a Predictive Factor During Weaning Process
Brief Title: PPI in Weaning Prediction
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, veysel Dinç, Assist. Prof., Gaziosmanpasa Research and Education Hospital
Other Study IDs: Gaziosmanpaşa TREH, VD
Record Dates: First submitted 2025-05-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Perfusion Index; Weaning of Mechanical Ventilation; ICU
Keywords: perfusion index; weaning; ıcu

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients were monitored for reentubation for 48 hours. — patients were monitored for reentubation for 48 hours.
Other: weaning group — patients were monitored for reentubation for 48 hours.

SUMMARY:
The aim of this study is to evaluate the predictive role of the Peripheral Perfusion Index (PPI) in forecasting extubation success during the weaning process in intensive care unit (ICU) patients. The study will investigate the ability of PPI to predict extubation failure by comparing it with traditional weaning criteria, including the Rapid Shallow Breathing Index (RSBI), PaO₂/FiO₂ ratio, and respiratory rate.

DETAILED DESCRIPTION:
Study Protocol This prospective observational study will be conducted in the Anesthesia Intensive Care Unit of Istanbul Gaziosmanpaşa Training and Research Hospital (SUAM) between March 2025 and June 2025 following approval from the Ethics Committee. Written informed consent will be obtained from the patients' legal representatives prior to enrollment.

Readiness for weaning from mechanical ventilation will be evaluated by the same attending intensivist throughout the study, in accordance with the local protocol. Criteria for readiness include resolution of the underlying cause of mechanical ventilation, ability to tolerate temporary discontinuation of mechanical ventilation, absence of frequent endotracheal suctioning needs, adequate oxygenation (PaO₂ > 60 mmHg with FiO₂ ≤ 0.5 and PEEP ≤ 8 cmH₂O), acceptable pH and PaCO₂ based on the patient's baseline respiratory condition, and stable cardiovascular status. In patients at high risk for upper airway edema, a cuff leak test will be performed by the intensivist.

The spontaneous breathing trial (SBT) will be performed using the Pressure Support (PS) mode with 5 cmH₂O PS and 5 cmH₂O PEEP. After 30 minutes, weaning parameters will be reassessed and the intensivist will make the extubation decision.

SBT failure will be defined by the presence of one or more of the following criteria: altered mental status, respiratory rate > 35 breaths/min, RSBI > 105, signs of increased respiratory effort (use of accessory muscles, thoracoabdominal asynchrony, intercostal retractions), SpO₂ < 90% or PaO₂ < 60 mmHg on FiO₂ of 0.4, or hemodynamic instability (heart rate > 140 bpm, systolic blood pressure > 180 mmHg or < 90 mmHg, or a change in either > 20% from baseline).

Patients with successful SBT will be extubated and monitored for 48 hours for the need for reintubation. Supplemental oxygen will be provided via a simple oxygen mask (4-6 L/min) to maintain SpO₂ > 92%.

The primary outcome is the ability of the Peripheral Perfusion Index (PPI) measured 1 hour after extubation to predict extubation failure within 48 hours.

The secondary outcomes include the predictive ability of PPI measured at the beginning of SBT, at 15 minutes, at the end of SBT, and 2 hours after extubation in identifying patients who will require reintubation within 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been on mechanical ventilation for at least 48 hours
* Patients over 18 years of age who are planned to undergo extubation following a spontaneous breathing trial (SBT)
* Patients or their legal representatives who provide informed consent to participate in the study

Exclusion Criteria:

* Patients for whom extubation is not planned due to hemodynamic instability
* Patients with peripheral vascular disease or a history of hand surgery
* Patients who die or cannot be followed up during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been on mechanical ventilation for at least 48 hours and Patients over 18 years of age who are planned to undergo extubation following a spontaneous breathing trial (SBT) Patients or their legal representatives who provide informed consent to participate in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
• The ability of Peripheric Perfusion Index(PPI) measured 1 hour after extubation to predict extubation failure within 48 hours following extubation. | 48 hours

SECONDARY OUTCOMES:
• The predictive power of Peripheric Perfusion Index(PPI) measured at the beginning of the spontaneous breathing trial (SBT), at the 15th minute, at the end of SBT, and 2 hours after extubation in determining extubation success. | 3 hours
• Correlation of Peripheric Perfusion Index(PPI) measurements between cardiac patients(Patients with at least one diagnosis of cardiac disease) and non-cardiac patients. | 48 hours
Changes in Peripheric Perfusion Index(PPI) values in patients who experience spontaneous breathing trial(SBT) failure. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No